CLINICAL TRIAL: NCT05288283
Title: A Randomized, Double-blind, Placebo-controlled, Multisite, Phase 3 Study to Investigate the Efficacy and Safety of Cannabidiol Oral Solution (GWP42003-P) in Children and Adolescents With Epilepsy With Myoclonic-Atonic Seizures
Brief Title: Efficacy and Safety of GWP42003-P Oral Solution in Children With Epilepsy With Myoclonic-atonic Seizures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to a business decision.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWEP20238
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Seizures Associated With EMAS
Keywords: Epilepsy; Seizures; Epilepsy with Myoclonic-Atonic Seizures (EMAS); Myoclonic-Atonic Epilepsy; Doose syndrome; Myoclonic-Astatic epilepsy (MAE); Children; Cannabidiol (CBD); GWP42003-P
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsies, Myoclonic | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GWP42003-P (Experimental): Participants will be initiated on a dose of GWP42003-P 2.5 milligrams per kilogram (mg/kg) twice a day (BID) (5 mg/kg/day); after 1 week, the dose will be increased to 5 mg/kg BID (10 mg/kg/day). Dose escalation up to a maximum daily dosage of 20 mg/kg/day (in increments of 5 mg/kg/day [2.5 mg/kg BID] no more rapidly than every 7 days) may occur after Day 15 based on the investigator's assessment of efficacy, safety and tolerability.
  Interventions: Drug: GWP42003-P
- Placebo (Placebo Comparator): Participants will receive the matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GWP42003-P — oral solution
  Other Names: EPIDIOLEX; Cannabidiol; Cannabidiol oral solution (CBD-OS)
  Arms: GWP42003-P
Drug: Placebo — oral solution
  Arms: Placebo

SUMMARY:
The primary aim of Part A of the study to assess the efficacy and tolerability of GWP42003-P compared to placebo as an adjunctive treatment for children with Epilepsy with myoclonic-atonic seizures (EMAS) -associated seizures.

Part B of this study will be conducted to evaluate the long-term safety and tolerability of GWP42003-P in participants with EMAS.

DETAILED DESCRIPTION:
The duration of study participation in Part A will be approximately 26 weeks, which includes a 1- to 3-week Screening Period, 4-week Baseline Observation Period, 14-week Dose Optimization Treatment Period, 10-day Taper Period, and a Safety Follow-up Period (4 weeks after end of taper visit). Participants will be randomized centrally in a 1:1 ratio to receive either GWP42003-P or matching placebo. Randomization will be stratified by clobazam use (on/off) and age of seizure onset (3 years of age and younger or older than 3 years of age). Upon completion of the double-blind phase (Part A), participants will have an option to continue in a 54-week open-label extension (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Participant has a current diagnosis of epilepsy with myoclonic-atonic seizures (EMAS), also known as Doose syndrome, myoclonic-astatic epilepsy, or myoclonic-atonic epilepsy, consistent with the International League Against Epilepsy (ILAE) guidelines. Presence of myoclonic-atonic seizures is mandatory to support a diagnosis of EMAS as determined by medical history and independent approval by The Epilepsy Study Consortium (TESC).
* Participant's initial seizure onset occurred from ≥ 6 months to < 6 years of age, with normal or mildly impaired/delayed neurodevelopment reported prior to onset of seizures. During the first year of seizure onset, the majority of seizures experienced by the participant were myoclonic-atonic seizures or generalized tonic-clonic seizures as determined by medical history.
* Participant is currently treated with one or more antiepileptic drug (AED) on a stable regimen (≥ 28 days prior to starting the baseline period [Part A Visit 2]) or on a stable ketogenic diet (≥ 3 months prior to starting the baseline period [Part A Visit 2]) and no changes to treatment are planned for the duration of the study.
* Participant is refractory to anticonvulsant medication and failed at least 1 AED (e.g., valproic acid, clobazam, clonazepam, and levetiracetam) at therapeutic doses.
* Participant is able to provide a historical electroencephalogram (EEG) report, which was performed within 12 months of Screening (Part A Visit 1), or is willing to complete an EEG at Screening (Part A Visit 1), that confirms a 3 to 6 Hertz (Hz) generalized spike-and-slow-wave or polyspike-and-slow-wave pattern.
* Contraceptive use by male and female participants should be consistent with Clinical Trial Facilitation Group (CTFG) guidelines and any applicable local regulations regarding the methods of contraception for those participating in clinical studies.

  1. Fertile male participants with partners of childbearing potential (CBP) must be willing to use a male barrier method of contraception in addition to a second method of acceptable contraception used by their female of CBP partners, from the time of Screening (Part A Visit 1) until 3 months after the follow-up visit.
  2. Female participants of CBP will not be pregnant or lactating and have a confirmed negative highly sensitive serum pregnancy test at Screening (Part A Visit 1).
  3. Female participants must also have a confirmed negative urine pregnancy test prior to receiving their first dose of blinded investigational medicinal product (IMP) at Part A Visit 3.
  4. Female participants who are continuing to Part B must have a confirmed negative urine pregnancy test prior to receiving their first dose of open-label GWP42003-P at Part B Visit 1.
  5. Female participants of CBP must be willing to use a highly effective method of contraception from the time of signing the Informed Consent Form (ICF) until 3 months after the follow-up visit.
* Participant or participant's caregiver(s) (according to local laws) is/are willing and able to give signed informed consent for participation in the study including compliance with the requirements and restrictions listed in the ICF and in the protocol.
* Participant's caregiver(s) are willing to allow the responsible authorities to be notified of participation in the study, if mandated by local law.
* Participant's caregiver completes at least 89% of Seizure eDiary entries during the first 28 days of the Baseline period (≥ 25 days of entries).

Part B only:

* Has completed Part A of this study
* Was compliant with all requirements of Part A (e.g., dosing, seizure eDiary, visits/procedures), in the judgement of the investigator and sponsor

Exclusion Criteria:

* Has a history of psychogenic non-epileptic seizures that confounds the assessment of the primary efficacy measure
* Has clinically significant unstable medical condition(s), other than EMAS
* Has a clinically significant illness in the 28 days prior to Screening (Visit 1) or randomization (Part A Visit 3), other than epilepsy, which in the opinion of the investigator could affect seizure frequency
* Has presence of focal seizures or persistent focal epileptiform discharges on EEG
* Has a history of infantile spasms
* Has moderate to severe neurocognitive and/or developmental delay prior to seizure onset
* Has a progressive neurological condition
* Has known or suspected hypersensitivity to cannabinoids or any of the excipients of GWP42003-P such as sesame oil
* Is unwilling or unable to remain stable on concurrent AEDs throughout the study.
* Has, in the opinion of the investigator, clinically significant abnormalities in the electrocardiogram (ECG) measured at Screening (Part A Visit 1), or any concurrent cardiovascular conditions, which will interfere with the ability to read their ECGs
* Has significantly impaired hepatic function at the Screening visit (Visit 1) or prior to dosing, defined as any of the following:

  1. alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 × upper limit of normal (ULN);
  2. total bilirubin (TBL) (serum) ≥ 2 × ULN or International Normalized Ratio (INR) > 1.5 (TBL ≥ 2 × ULN exclusion will not apply for participants diagnosed with Gilbert's disease);
  3. serum ALT or AST ≥ 3 × ULN with the presence of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%);
  4. elevated ALT or AST at Screening (Part A Visit 1), should be discussed with the medical monitor prior to Randomization (Part A Visit 3); the medical monitor may allow for a confirmatory re-draw prior to randomization.

This criterion can only be confirmed once the laboratory results are available.

* Has clinically significant impaired renal function at Screening (Part A Visit 1), as evidenced by an estimated creatinine clearance lower than 60 milliliters per minute (mL/min)
* Is a female participant of CBP, who is pregnant (positive pregnancy test), lactating or planning pregnancy during the course of the study and for 3 months thereafter
* Participant has any known or suspected history of alcohol or substance abuse
* Any clinically significant abnormalities identified following a physical examination or laboratory assessments of the participant that, in the opinion of the investigator, would jeopardize the safety of the participant if they take part in the study
* Participant has any other clinically significant disease or disorder which, in the opinion of the investigator, may either put the participant, other participants, or site staff at risk because of participation in the study, may influence the result of the study, or may affect the participant's ability to take part in the study
* Has a change in anticonvulsant therapies within 28 days of starting the baseline period (Part A Visit 2), including AEDs or settings on vagal nerve stimulator
* Has any planned clinical interventions or intends to change any or all medications that may impact seizures during the study
* Has been treated with a general anesthetic in the 28 days prior to screening (Part A Visit 1) or randomization (Part A Visit 3 [Week 0])
* Has undergone surgery for epilepsy in the 6 months prior to Screening (Part A Visit 1)
* Is being considered for epilepsy surgery or any procedure involving general anesthesia during the study
* Has initiated a ketogenic diet within 3 months prior to the Baseline period (Part A Visit 2). Participants who are stable on a ketogenic diet for ≥ 3 months and willing to remain on a stable epilepsy dietary therapy (e.g., ketogenic diet, Atkins diet, low glycemic index diet) during the study, are eligible for inclusion.
* Has initiated felbamate within 12 months prior to screening (Part A Visit 1). Participants who are stable on a felbamate for ≥ 12 months are eligible for inclusion.
* Is currently being treated with or had previously (within 3 months prior to screening [Part A Visit 1] received intravenous immunoglobulin treatment or plasma exchange for the treatment of seizures
* Has participated in a clinical study involving administration of an IMP (new chemical entity) or medical device (e.g., vagal nerve stimulator) within 1 month prior to screening (Part A Visit 1)
* Have previously been randomized, completed, or withdrawn from this study
* Is currently using a drug of abuse or current non-prescribed use of any prescription drug
* Is currently using or has used recreational or medicinal cannabis, cannabinoid-based medications, products, or supplements (botanical or synthetic) within 28 days prior to screening (Part A Visit 1).
* Mother (if breastfeeding the participant) is currently using or has used recreational or medicinal cannabis, cannabinoid-based medications, products, or supplements (botanical or synthetic) within 28 days of screening (Part A Visit 1).
* Has any history of suicidal behavior or serious suicidal ideation, defined as Category 4 or greater on the Columbia Suicide Severity Rating Scale (C-SSRS) at any visit prior to dosing with IMP. This criterion applies only to participants 4 to 18 years of age.
* Is unwilling or unable to comply with all study requirements, including accurate eDiary completion
* Participants who, in the opinion of the investigator (or designee), should not participate in this study
* Has travel planned outside their country of residence during the study, unless the participant has confirmation that the IMP is permitted in the destination country and all stops along the way

Part B only:

* Has significantly impaired hepatic function at Part A Visit 9, defined as any of the following:

  1. ALT or AST > 5 × ULN;
  2. TBL (serum) ≥ 2 × ULN or INR > 1.5 (TBL ≥ 2 × ULN exclusion will not apply for participants diagnosed with Gilbert's disease.
  3. Serum ALT or AST ≥ 3 × ULN with the presence of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%). The medical monitor may allow for a confirmatory redraw prior to rollover.
* Meets any exclusion criteria at Part B Visit 1

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (10):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of California Davis Health, Sacramento, California
  - Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Wake Forest Baptist Health Sciences, Department of Neurology, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center - TS Clinic, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell's Children's Hospital, Austin, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Italy (4):
  - Azienda Ospedaliero Universitaria Ospedale Pediatrico Meyer, Florence
  - Istituto Giannina Gaslini-Ospedale Pediatrico IRCCS, Genova
  - IRCCS Fondazione Istituto Neurologico Nazionale D. Mondino Pavia, Pavia
  - UOC Neuropsichiatria Infantile AOUI Verona, Verona

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened for enrollment at 14 activated sites: 10 in the USA and 4 in Italy.
Pre-assignment Details: A total of 3 participants were enrolled in Part A of the study. One participant was a screen failure, and 2 underwent randomization. Study was terminated prior to Part B.
Groups:
- GWP42003-P: Participants who received a dose escalation of GWP42003-P twice a day (BID) orally.
- Placebo: Participants who received the matching placebo.
Period: Overall Study
Arm/Group | GWP42003-P | Placebo
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Study Terminated Early | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GWP42003-P | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percent Change From Baseline in Epilepsy With Myoclonic-atonic Seizures (EMAS) Associated Seizure Frequency (Myoclonic-atonic, Atonic, Tonic, Clonic, or Tonic-clonic) Over the 14-week Treatment Period
Time Frame: Baseline; up to 14 weeks
Population: No data collected, as the study was terminated before this endpoint was analyzed.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Part B: Number of Participants With Treatment-emergent Adverse Events
Time Frame: up to Week 54
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Part B: Number of Participants With Clinically Significant Vital Sign Values
Time Frame: up to Week 50
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Part B: Number of Participants With Clinically Significant Physical Examination Values
Time Frame: up to Week 48
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Part B: Number of Participants With Clinically Significant 12-lead Electrocardiogram (ECG) Values
Time Frame: up to Week 48
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Part B: Number of Participants With Clinically Significant Laboratory Test Values
Time Frame: up to Week 48
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Part B: Number of Participants With Changes in Tanner Staging
Time Frame: up to Week 48
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Part B: Number of Participants With a Change in Columbia-Suicide Severity Rating Scale (C-SSRS) Ideation Scores
Time Frame: up to Week 54
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Part B: Number of Participants With a Change in the Number of Suicide Attempts Per C-SSRS Scores
Time Frame: up to Week 54
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Part A: Number of Participants Who Achieve ≥ 50% Reduction From Baseline in EMAS-associated Seizures Over the 14-week Treatment Period
Time Frame: Baseline; up to 14 weeks
Population: No data collected, as the study was terminated before this endpoint was analyzed.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Part A: Total Seizure Frequency Over the 14-week Treatment Period
Time Frame: Baseline; up to 14 weeks
Population: No data collected, as the study was terminated before this endpoint was analyzed.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Part A: Caregiver Global Impression of Change (CGIC) Score at Week 14
Time Frame: Week 14
Population: No data collected, as the study was terminated before this endpoint was analyzed.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Part A: Physician Global Impression of Change (PGIC) Score at Week 14
Time Frame: Week 14
Population: No data collected, as the study was terminated before this endpoint was analyzed.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Part A: Number of Participants Who Achieve ≥ 25%, ≥ 50%, ≥ 75%, and 100% Reduction From Baseline in Total Seizures Over the 14-week Treatment Period
Time Frame: Baseline; up to 14 weeks
Population: No data collected, as the study was terminated before this endpoint was analyzed.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Part A: Change From Baseline in the Number of EMAS-associated Seizure-free Days Over the 14-week Treatment Period
Time Frame: Baseline; up to 14 weeks
Population: No data collected, as the study was terminated before this endpoint was analyzed.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Part A: Number of Participants With at Least 25% and 50% Reduction From Baseline in the Number of Days Per Week With Myoclonic Seizures During the 14-week Treatment Period
Time Frame: Baseline; up to 14 weeks
Population: No data collected, as the study was terminated before this endpoint was analyzed.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Part A: Time to Baseline Seizure Frequency
Time Frame: up to 14 weeks
Population: No data collected, as the study was terminated before this endpoint was analyzed.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Part A: Number of Participants With Treatment-emergent Adverse Events
Description: A TEAE is an adverse event that started or worsened in severity or seriousness following the first dose of the investigational medicinal product.
Time Frame: From the time of informed consent signing up to 27 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

19. Secondary Outcome: Part A: Number of Participants With Clinically Significant Laboratory Test Values
Time Frame: up to 27 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

20. Secondary Outcome: Part A: Number of Participants With Clinically Significant Vital Sign Values
Time Frame: up to 27 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

21. Secondary Outcome: Part A: Number of Participants With Clinically Significant Physical Examination Values
Time Frame: up to 27 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

22. Secondary Outcome: Part A: Number of Participants With Clinically Significant 12-lead ECG Values
Time Frame: up to 27 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

23. Secondary Outcome: Part A: Number of Participants With Changes in Tanner Staging
Time Frame: up to Day 99
Population: No data collected, as the study was terminated before this endpoint was analyzed.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Part A: Number of Participants With a Change in C-SSRS Ideation Scores
Time Frame: up to 27 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

25. Secondary Outcome: Part A: Number of Participants With a Change in the Number of Suicide Attempts Per C-SSRS Scores
Time Frame: up to 27 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

26. Secondary Outcome: Part B: Percent Change From Baseline in EMAS-associated Seizure Frequency (Myoclonic-atonic, Atonic, Tonic, Clonic, or Tonic-clonic) Over the 48-week Open-label Treatment Period
Time Frame: Baseline; up to 48 weeks
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Part B: Number of Participants Achieving ≥50% Reduction From Baseline in EMAS-associated Seizures Over the 48-week Open-label Treatment Period
Time Frame: Baseline; up to 48 weeks
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Part B: Total Seizure Frequency Over the 48-week Open-label Treatment Period
Time Frame: up to Week 48
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Part B: CGIC Score at Weeks 14, 24, and 48
Time Frame: Weeks 14, 24, and 48
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Part B: PGIC Score at Weeks 14, 24, and 48
Time Frame: Weeks 14, 24, and 48
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Part B: Number of Participants Who Achieve ≥ 25%, ≥ 50%, ≥ 75%, and 100% Reduction From Baseline in Total Seizures Over the 48-week Open-label Treatment Period
Time Frame: Baseline; up to 48 weeks
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Part B: Change From Baseline in the Number of EMAS-associated Seizure-free Days Over the 48-week Open-label Treatment Period
Time Frame: Baseline; up to 48 weeks
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Part B: Number of Participants With at Least 25% and 50% Reduction From Baseline in the Number of Days Per Week With Myoclonic Seizures During the 48-week Open-label Treatment Period
Time Frame: Baseline; up to 48 weeks
Population: Not data was collected, as the study was terminated prior to part B.
Arm/Group | GWP42003-P | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All treatment-emergent adverse events (TEAE) were collected from signing the informed consent up to approximately 27 weeks. No participants entered the open-label extension phase due to study termination.
Description: A TEAE is an adverse event that started or worsened in severity or seriousness following the first dose of the investigational medicinal product.
Arm/Group | GWP42003-P | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P (N=1) | Placebo (N=1)
Gastroenteritis viral (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P (N=1) | Placebo (N=1)
Irritability (Psychiatric disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Blood triglycerides (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT05288283/Prot_SAP_003.pdf